CLINICAL TRIAL: NCT06625749
Title: Early Feasibility Study to Evaluate the Safety and Effectiveness of the AccuraSee™ IOPCL for Secondary Implantation in the Capsular Bag to Improve Near and/or Intermediate Vision Following Previous Cataract Surgery
Brief Title: Evaluate the Safety and Effectiveness of the AccuraSee™ IOPCL for Secondary Implantation in the Capsular Bag to Improve Near and/or Intermediate Vision Following Previous Cataract Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OnPoint Vision Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIIPCL-022R
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Refractive Surgery; Refractive Error - Myopia
Keywords: IOPCL; Refractive error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AccuraSee™ intraocular pseudophakic capsular lens (IOPCL) (Experimental)
  Interventions: Device: Accurasee™ IOPCL

INTERVENTIONS:
Device: Accurasee™ IOPCL — Intraocular pseudophakic capsular lens (IOPCL)

SUMMARY:
This is a study to evaluate the safety and effectiveness of the AccuraSee™ intraocular pseudophakic capsular lens (IOPCL) to improve near and/or intermediate vision following previous cataract surgery.

DETAILED DESCRIPTION:
The objective of this study is to provide preliminary evidence of the safety and efficacy of the AccuraSee intraocular pseudophakic capsular lens (IOPCL) in qualified subjects previously implanted with an Alcon monofocal intraocular lens model SN60WF, SA60WF, or SA60AT, Johnson and Johnson model ZCB00, or Zeiss model CT LUCIA 602 who desire near vision of 20/32 or better via a myopic shift in the eye to be treated.

ELIGIBILITY:
Inclusion Criteria:

All ocular eligibility criteria refer to the study (non-dominant) eye only unless otherwise noted.

1. Subjects aged 22 years and older.
2. Subjects who have had cataract surgery with an Alcon monofocal intraocular lens model SN60WF, SA60WF, or SA60AT (with a lens power from 10.0D to 30.0D), or Johnson and Johnson monofocal lens model ZCB00 (with a lens power from 10.0D to 26.0D), or Zeiss monofocal lens model CT LUCIA 602 (with a lens power from 10.0D to 19.0D) clearly evidenced by photographic documentation with one of the following: patient medical record, clinic chart with labeling attached, surgical record with labeling attached, or patient identification card with make, model, power and serial number.
3. Subjects who have had cataract surgery at least 6 months from the planned date of IOPCL surgery.
4. Subjects who require a reading add of +1.50 to +2.50 to achieve an BCNVA of 20/32 or better.
5. Subjects with uncorrected near visual acuity (UCNVA) 20/50 or worse.
6. Subjects with best corrected distance visual acuity (BCDVA) 20/25 or better in both eyes.
7. Subjects with uncorrected distance visual acuity (UCDVA) 20/25 or better in fellow eye.
8. Subjects with best corrected near visual acuity (BCNVA) 20/32 or better.
9. Subjects with a manifest refraction spherical equivalent (MRSE) in the study eye between +0.25D and +1.50D.
10. Subjects with <1D of refractive cylinder determined by keratometry readings.
11. Subjects with a minimum endothelial cell count of 1800 cells/mm2.
12. Subjects with a tear break up time (TBUT) ≥ 7 seconds.
13. Subjects with a documented monovision tolerance, or who have successfully completed a 1-week contact lens trial prior to implantation with the IOPCL.
14. For subjects who are contact lens wearers, discontinuation of lens usage prior to the preoperative visit (at least 2 weeks for subjects using soft contact lenses and at least 3 weeks for hard or rigid gas permeable (RGP) lenses) except as required to test monovision acceptance.
15. For subjects who are contact lens wearers, two central keratometry readings with regular mires and two manifest refractions taken at least one week apart (keratometry values must not differ by more than ±0.50D in either principal meridian in the eye to be treated).
16. Subjects able to comprehend and sign a statement of informed consent.
17. Subjects willing and able to complete all required postoperative visits.
18. Subjects willing to abstain from pursuing any other refractive surgery for the duration of the study.

Exclusion Criteria:

1. Subjects who have had cataract surgery with other than a monofocal posterior chamber intraocular lens (PCIOL).
2. Subjects who have had previous laser refractive surgery.
3. Subjects who have had cataract surgery with an Alcon monofocal intraocular lens model SN60WF, SA60WF, or SA60AT (with a lens power below 10.0D or greater than 30.0D), or Johnson and Johnson monofocal intraocular lens model ZCB00 (with a lens power below 10.0D or greater than 26.0D) or Zeiss monofocal lens model CT LUCIA 602 (with a lens power below 10.0D or greater than 19.0D).
4. Subjects who were treated with a PCIOL in a manner that is not consistent with the labeling, contraindications, or indications for use statement.
5. Subjects whose continuous curvilinear capsulorhexis is less than 4.5 mm or more than 6.0 mm in size at the time of the preoperative visit.
6. Subjects who have had a Nd:YAG capsulotomy less than 1 month prior to the planned date of the IOPCL surgery.
7. Subjects with a mesopic non-dilated pupil of greater than 5.5mm.
8. Subjects with a mesopic dilated pupil of less than 7.0 mm.
9. Subjects who have 1D or more of refractive cylinder determined by keratometry readings.
10. Subjects who had cataract surgery less than 6 months from the planned date of the IOPCL surgery.
11. Subjects whose PCIOL is substantially decentered (> 1.0 mm).
12. Subjects with anterior capsule fibrosis and phimosis that, in the opinion of the investigator, may confound the outcome or increase the risk to the subject (e.g., excessive capsule contraction potentially obstructing the visual axis or causing late secondary complications to the PCIOL such as pseudophacodenesis and IOL tilt, decentration, or dislocation due to zonular laxity, weakness or dehiscence).
13. Subjects with capsular instability.
14. Subjects with an anterior capsular defect.
15. Subjects with posterior capsular defect < 0.5 mm from the edge of the existing IOL (caused by Nd:YAG capsulotomy).
16. Subjects with a tear or rent in the anterior or posterior capsule.
17. Subjects with any corneal pathology that is either progressive or sufficient to reduce BCDVA to 20/25 or worse.
18. Subjects with any corneal abnormality, other than regular corneal astigmatism, that prevents accurate assessment of fluorescein tear break up time or, in the opinion of the investigator, would confound the outcome(s) of the study.
19. Subjects with active moderate to severe meibomian gland dysfunction.
20. Subjects with clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy).
21. Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that would reduce BCDVA to 20/25 or worse.
22. Subjects with recurrent severe anterior or posterior segment inflammation of unknown etiology.
23. Subjects with microphthalmos.
24. Subjects with previous retinal detachment.
25. Subjects with diabetic retinopathy.
26. Subjects with iris neovascularization.
27. Subjects with a history of steroid-responsive rise in intraocular pressure (IOP), uncontrolled glaucoma or preoperative IOP >21 mmHg.
28. Subjects with amblyopia in either eye.
29. Subjects who have current or historical significant binocular muscle imbalances or intermittent tropias and/or fail the cover test.
30. Subjects who fail to demonstrate normal perception at near (33 cm) on the Worth 4 Dot Binocular Test for binocular function (using best corrected visual acuity).
31. Subjects who fail to demonstrate at least gross stereopsis (i.e., pinching fly's wings in front of test booklet) with best corrected visual acuity on the Titmus Stereo Test (at near).
32. Subjects with a fundus not visible.
33. Subjects with aniridia.
34. Subjects with optic nerve atrophy.
35. Subjects with damaged or incomplete zonules.
36. Subjects with inadequate anterior leaflet coverage of the PCIOL (defined as less than 0.5 mm of anterior leaflet of capsule above where the haptics will reside).
37. Subjects with damage to the PCIOL.
38. Subjects with a known history of pseudoexfoliation, or pseudoexfoliation diagnosed at the preoperative visit or prior to IOPCL implantation.
39. Subjects with acute, chronic or uncontrolled systemic or ocular disease that in the opinion of the investigator would increase the operative risk or confound the outcome(s) of the study.
40. Subjects taking medications that, in the opinion of the investigator, may confound the outcome or increase the risk to the subject (tamsulosin hydrochloride (Flomax)) or taking other medications with similar side effects (floppy iris syndrome).
41. Subjects participating in any other ophthalmic drug or device trial during the time of this investigation.
42. Subjects who are pregnant or nursing women; or women of child bearing age not using medically acceptable contraceptives.
43. Subjects with certain occupational and environmental visual demands (i.e. piloting an airplane, working on and operating dangerous machinery) in the opinion of the investigator would increase the post-operative risk.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in uncorrected near visual acuity (UCNVA) at 40 cm/16 inches | 12 months
  Improvement in uncorrected near visual acuity (UCNVA) (at 40 cm/16 inches) at 12 months postoperatively. At least 75% of treated eyes should achieve an uncorrected near visual acuity (UCNVA) of 20/32 or better.

OTHER OUTCOMES:
Improvement in uncorrected intermediate visual acuity (UCIVA) (at 66 cm/26 inches) | 12 months
  Improvement in uncorrected intermediate visual acuity (UCIVA) at 66 cm/26 inches at 12 months postoperatively. At least 75% of treated eyes should achieve a UCIVA of 20/40 or better.
Preservation of best corrected distance visual acuity (BCDVA) | 12 Months
  Proportion of eyes (< 5%) that lose two or more lines of best corrected distance visual acuity (BCDVA) (≥ 10 letters on the Early Treatment for Diabetic Retinopathy Study [ETDRS] chart).
Successful delivery of the intraocular pseudophakic capsular lens (IOPCL) | Postoperatively from 7-14 days visit through 12 months visit
  Successful delivery of the intraocular pseudophakic capsular lens (IOPCL) (defined as no capsular tear, no visible damage to either the posterior chamber intraocular lens [PCIOL] or the IOPCL, and adequate leaflet coverage of all IOPCL haptic tabs [≥ 0.5 mm of anterior leaflet of capsule above where the haptics reside]).
PCIOL Long-term adherence and positional stability (tilt) | Postoperatively from 30-60 days visit through 12 months visit
  Minimal tilt of the posterior chamber intraocular lens (PCIOL) confirmed via Anterion® AS-OCT (defined as ≤ 10 degrees between the postoperative tilt of the PCIOL and the pre-operative tilt of the PCIOL).
Intraocular Pseudophakic Capsular Lens (IOPCL) Long-term adherence and positional stability (tilt) | Postoperatively from 30-60 days visit through 12 months visit
  Minimal tilt of the intraocular pseudophakic capsular lens (IOPCL) (using the posterior chamber intraocular lens [PCIOL] as a reference point) confirmed via Anterion® AS-OCT (defined as ≤ 10 degrees between the post-operative tilt of the PCIOL and the postoperative tilt of the IOPCL).
PCIOL/IOPCL Complex Long-term adherence and positional stability (decentration) | Postoperatively starting at 7-14 days through 12 months
  Decentration of the posterior chamber intraocular lens/intraocular pseudophakic capsular lens (PCIOL/IOPCL complex) (defined as uniform exposed area of the PCIOL outside of the IOPCL at the vertical and horizontal meridians between ≥ 0.5 mm and ≤ 1.0 mm.
Intraoperative and postoperative adverse events | Intraoperative and Postoperative through 12 months
  Characterization and incidence of cumulative and persistent intraoperative and post-operative adverse events.
Secondary Surgical Interventions (SSIs) | Postoperative through 12 months
  Incidence of secondary surgical interventions (SSIs) (e.g., removal of interlenticular opacity, repositioning of intraocular pseudophakic capsular lens [IOPCL], explant of IOPCL, repositioning of posterior chamber intraocular lens [PCIOL]) (excluding neodymium-doped yttrium aluminum garnet [Nd:YAG] treatments for posterior capsule opacification (PCO).
Endothelial Cell Counts | Postoperatively beginning with 120-180 days through 12 months
  Endothelial Cell Counts (mean loss, minimum, maximum, and quartiles of endothelial cell density [ECD] loss)
  * Percent of eyes that lose 20% or more ECD
  * Percent of eyes that lose 25% or more ECD
  * Percent of eyes that lose 30% or more ECD

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Vision Partners, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No